CLINICAL TRIAL: NCT03642899
Title: Study of Peripapillary Vasculature With OCT-angiography in Arteritic and Non Arteritic Anterior Ischemic Neuropathy After Oedema Disappearance
Brief Title: OCT Angiography in Arteritic and Non Arteritic Anterior Ischemic Neuropathy
Acronym: NOIA
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NOIA
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Neuropathy, Optic
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with anterior ischaemic optic neuropathy: estimation of best visual acuity, fondus, measurement of retinal nervous layer thickness, ganglionar cells layer thickness, and a macular and papillar OCT angiography during a consultation
- control group. Normal eyes: estimation of best visual acuity, fondus, measurement of retinal nervous layer thickness, ganglionar cells layer thickness, and a macular and papillar OCT angiography during a consultation

SUMMARY:
Anterior ischaemic optic neuropathy results from infarction of retrolaminar portion of the optic nerve head, caused by occlusion of the posterior ciliary artery. Non arteritic anterior ischaemic optic neuropathy affects more frequently people between 50 and 70 years of age, with vasculopathic risk factors. Arteritic anterior ischaemic optic neuropathy is caused by the Horton disease, affects an older population and is an ophthalmologic emergency because of the bilateralisation's risk.

The aim of this study is to compare the peripapillar vascular density of anterior ischaemic optic neuropathy eyes (arteritic and non arteritic) with normal eyes after the disappearance of the papillar edema, with oCT-angiography.

The investigators will include patients with anterior ischaemic optic neuropathy and normal patients. For each participant, the investigators will estimate the best visual acuity, intra-ocular pressure, make a fondus, measurement of retinal nervous layer thickness, ganglionar cells layer thickness, and a macular and papillar OCT angiography during a consultation (duration 30 min).

The investigators will be able to know if

* there is a modification of the peripapillary vascularisation subsequent to the occlusion of the posterior ciliary artery
* there is a difference between arteritic and non arteritic anterior ischaemic optic neuropathy,
* there is a repercussion of the neuropathy on the retinal layers,
* there is a difference in peripapillar vascularisation by age.

DETAILED DESCRIPTION:
Anterior ischaemic optic neuropathy results from infarction of retrolaminar portion of the optic nerve head, caused by occlusion of the posterior ciliary artery. Non arteritic anterior ischaemic optic neuropathy affects more frequently people between 50 and 70 years of age, with vasculopathic risk factors. Arteritic anterior ischaemic optic neuropathy is caused by the Horton disease, affects an older population and is an ophthalmologic emergency because of the bilateralisation's risk.

The aim of this study is to compare the peripapillar vascular density of anterior ischaemic optic neuropathy eyes (arteritic and non arteritic) with normal eyes after the disappearance of the papillar edema, with oCT-angiography.

The investigators will include patients with anterior ischaemic optic neuropathy and normal patients. For each participant, the investigators will estimate the best visual acuity, intra-ocular pressure, make a fondus, measurement of retinal nervous layer thickness, ganglionar cells layer thickness, and a macular and papillar OCT angiography during a consultation (duration 30 min).

The investigators will be able to know if

* there is a modification of the peripapillary vascularisation subsequent to the occlusion of the posterior ciliary artery
* there is a difference between arteritic and non arteritic anterior ischaemic optic neuropathy,
* there is a repercussion of the neuropathy on the retinal layers,
* there is a difference in peripapillar vascularisation by age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arteritic or non-arteritic anterior ischemic optic neuropathy ,> 3 months or after disappearance of papillary edema
* Control subjects, with normal optic nerve and symmetrical appearance , without diagnosed glaucoma (intraocular tension lower than 21mmHg) and without antecedent of retinal or intraorbital pathology.
* Patient with cataract can be included, within the limits of the good acquisition of images.
* Free, without tutorship or curatorship or subordination
* Benefiting from a Social Security scheme or benefiting through a third party
* Giving their non-opposition, after clear and fair information on the study

Exclusion Criteria:

* with ocular or retinal pathology leading to irreversible visual impairment or macular involvement (strong myopia> 6 diopters, astigmatism> 3 diopters, retinitis pigmentosa, occlusion of the central artery of the retina or central vein of the retina , CRSC, diabetic retinopathy), or history of ocular or retinal surgery except cataract surgery.
* having an alteration of the optic nerve related to another pathology (NORB, glaucoma evolved with cup / disc> 0.7 or poorly balanced tension, optic neuritis),
* performing the exam impossible or poor image quality
* impossibility of giving one's non-opposition,
* not benefiting from a social security scheme or benefiting from it through a third person
* benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with arteritic or non-arteritic anterior ischemic optic neuropathy ,> 3 months or after disappearance of papillary edema
  * Control subjects, with normal optic nerve and symmetrical appearance
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
compare peripapillary vascular density in eyes with anterior ischaemic optic neuropathy and in normal eyes with OCT angiography | 10 minutes
  Measurement of vascular density by percentage of area occupied by peripapillary vessels in patients with anterior ischemic optic neuropathy and control subjects

SECONDARY OUTCOMES:
compare vascular microvascular density at the macular level with angio-OCT in patients with anterior ischemic optic neuropathy and control subjects | 10 minutes
  Measurement of macular microvascular density by percentage of the area occupied by the vessels in patients with anterior ischemic optic neuropathy and control subjects,
Compare Peripapillary and Macular Mirovascular Differences in Arteritic and Non-Arteritic anterior ischemic optic neuropathy Patients | 10 minutes
  Measurement of microvascularisation density and its abnormalities (dilatation, defect) on peripapillary angio-OCT images in group with an arteritic optic neuropathy compared to patients with non-arteritic optic neuropathy
compare the microvascular density of the 2 optic discs in the same patient : with optic neuropathy and the healthy disc | 10 minutes
  Measurement of peripapillary microvascular density in the eye with anterior ischemic optic neuropathy and healthy contralateral eye in the same patient
compare the thickness of the peripapillary retinal nerve fibers and the thickness of the ganglionar complex layer in patients with anterior ischemic optic neuropathy and control group | 5 minutes
  Measurement of retinal nerve fiber thickness (RNFL), and thickness of ganglionic complex layer (GCC) with OCT in 2 groups
Compare peripapillary and macular microvascular density by age and by sex | 10 minutes
  Measurement of macular and peripapillary microvascular density on angio-OCT images for comparison between different age groups

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

REFERENCES:
- [Background] Balducci N, Morara M, Veronese C, Barboni P, Casadei NL, Savini G, Parisi V, Sadun AA, Ciardella A. Optical coherence tomography angiography in acute arteritic and non-arteritic anterior ischemic optic neuropathy. Graefes Arch Clin Exp Ophthalmol. 2017 Nov;255(11):2255-2261. doi: 10.1007/s00417-017-3774-y. Epub 2017 Aug 31. PMID 28861697
- [Background] Berry S, Lin WV, Sadaka A, Lee AG. Nonarteritic anterior ischemic optic neuropathy: cause, effect, and management. Eye Brain. 2017 Sep 27;9:23-28. doi: 10.2147/EB.S125311. eCollection 2017. PMID 29033621
- [Background] Gaier ED, Gilbert AL, Cestari DM, Miller JB. Optical coherence tomographic angiography identifies peripapillary microvascular dilation and focal non-perfusion in giant cell arteritis. Br J Ophthalmol. 2018 Aug;102(8):1141-1146. doi: 10.1136/bjophthalmol-2017-310718. Epub 2017 Nov 9. PMID 29122818
- [Background] Hata M, Oishi A, Muraoka Y, Miyamoto K, Kawai K, Yokota S, Fujimoto M, Miyata M, Yoshimura N. Structural and Functional Analyses in Nonarteritic Anterior Ischemic Optic Neuropathy: Optical Coherence Tomography Angiography Study. J Neuroophthalmol. 2017 Jun;37(2):140-148. doi: 10.1097/WNO.0000000000000470. PMID 27984351
- [Background] Ling JW, Yin X, Lu QY, Chen YY, Lu PR. Optical coherence tomography angiography of optic disc perfusion in non-arteritic anterior ischemic optic neuropathy. Int J Ophthalmol. 2017 Sep 18;10(9):1402-1406. doi: 10.18240/ijo.2017.09.12. eCollection 2017. PMID 28944200
- [Background] Liu CH, Kao LY, Sun MH, Wu WC, Chen HS. Retinal Vessel Density in Optical Coherence Tomography Angiography in Optic Atrophy after Nonarteritic Anterior Ischemic Optic Neuropathy. J Ophthalmol. 2017;2017:9632647. doi: 10.1155/2017/9632647. Epub 2017 Feb 19. PMID 28316838
- [Background] Moghimi S, Afzali M, Akbari M, Ebrahimi KB, Khodabande A, Yazdani-Abyaneh AR, Ghafouri SNH, Coh P, Okhravi S, Fard MA. Crowded optic nerve head evaluation with optical coherence tomography in anterior ischemic optic neuropathy. Eye (Lond). 2017 Aug;31(8):1191-1198. doi: 10.1038/eye.2017.56. Epub 2017 Apr 7. PMID 28387764
- [Background] Sharma S, Ang M, Najjar RP, Sng C, Cheung CY, Rukmini AV, Schmetterer L, Milea D. Optical coherence tomography angiography in acute non-arteritic anterior ischaemic optic neuropathy. Br J Ophthalmol. 2017 Aug;101(8):1045-1051. doi: 10.1136/bjophthalmol-2016-309245. Epub 2017 Jan 5. PMID 28057645
- [Background] Song Y, Min JY, Mao L, Gong YY. Microvasculature dropout detected by the optical coherence tomography angiography in nonarteritic anterior ischemic optic neuropathy. Lasers Surg Med. 2018 Mar;50(3):194-201. doi: 10.1002/lsm.22712. Epub 2017 Oct 7. PMID 28986994